CLINICAL TRIAL: NCT04390685
Title: Prevention of Breast Cancer-related Lymphedma With Tacrolimus
Acronym: BCRL-TACRO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Gustaf Jørgensen, Medical doctor, ph.d.-student., Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20180134; 2018-003416-50 (EudraCT Number)
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus ointment (Experimental): Apply whole arm, in a thin layer, once daily for one year
  Interventions: Drug: Tacrolimus ointment
- Control (No Intervention)

INTERVENTIONS:
Drug: Tacrolimus ointment — Treatment with tacrolimus ointment once daily for one year following axillary lymph node dissection
  Arms: Tacrolimus ointment

SUMMARY:
Breast cancer-related lymphedema is one of the most common and feared consequences of breast cancer treatment. Tacrolimus ointment may prevent lymphedema by inhibition of CD4+T cells.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Breast cancer with planned ALND
* postmenopausal or use of contraceptives
* good general health condition
* read and understand Danish

Exclusion Criteria:

* Pregnant, breastfeeding it wishing to conceive with the next year
* bilateral breast cancer
* known allergy to tacrolimus or macrolides
* known lymphedema
* other malignant disease apart from keratinocyte cancer
* in medical treatment for diabetes mellitus
* known psychiatric condition which may influence participation
* known renal or hepatic function

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Lymphedema | 1 year
  Arm size change >= 10% using water displacement

SECONDARY OUTCOMES:
Subjective changes assessed using the LYMPH-ICF (Lymphoedema Functioning, Disability and Health) questionaire | 1 year
  Subjective change of lymphedema assessed by questionnaire. Range: 0-100. 100 being the most bothered.
Subjective changes assessed using DASH (DISABILITIES OF THE ARM, SHOULDER AND HAND) questionaire | 1 year
  Subjective change of lymphedema assessed by questionnaire. Range: 1-5. 5 being the most bothered
Subjective changes assessed using SF-36 questionnaire (Short form-36) | 1 year
  Subjective change of lymphedema assessed by questionnaire. Range: 0-100. 0 being the most bothered
Change in L-DEX score using bioimpedance (Odense University Hospital Only). | 1 year
  Change in L-DEX score of lymphedema arm derived from bioimpedance. Higher values mean more fluid in the lymphedema arm compared to the healthy arm.
Change in lymph drainage. (Odense University Hospital Only). | 1 year
  Change in lymph drainage assessed by indocyanine-green lymphangiography

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Sydvestjysk Sygehus, Esbjerg
  - Department of Plastic and Reconstructive Surgery, Odense
  - Sygehus Lillebælt Vejle, Vejle

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Starting 1 year after publication
Access Criteria: Jens Ahm Sørensens review requests